CLINICAL TRIAL: NCT02410239
Title: MT2014-14 Intrathecal Administration of Mesenchymal Stem Cells (IT-MSC) for the Treatment of Advanced Cerebral Adrenoleukodystrophy (cALD)
Brief Title: MT2014-14 IT-MSC for Advanced Cerebral Adrenoleukodystrophy (cALD)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Research cancelled
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014LS018
Record Dates: First submitted 2015-03-27; First posted 2015-04-07 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Cerebral Adrenoleukodystrophy
Keywords: Cerebral Adrenoleukodystrophy; cALD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal Stem Cell (Experimental): Third party donor Mesenchymal Stem Cells (MSC) will be administered via intrathecal administration at the assigned dose on days 0, 7 and 14. Dose escalation will be guided by a fast track design. One patient is entered per dose level until a DLT is experienced. At that point, two additional patients will be enrolled at the same dose level. Dose levels will be 2.5 x 10e6 MSC/kg per dose, 5 x 10e6 MSC/kg per dose or 7.5 x 10e6 MSC/kg per dose.
  Interventions: Biological: Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Mesenchymal Stem Cells

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of mesenchymal stem cells (IT-MSC) in patients with active, advanced cerebral adrenoleukodystrophy (cALD).

DETAILED DESCRIPTION:
This is a single-institution dose escalation study to determine the maximum tolerated dose (MTD) of intrathecally administered allogeneic, 3rd party mesenchymal stem cells (IT-MSC) in patients with active, advanced cerebral adrenoleukodystrophy (cALD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 4 years at time of study enrollment
* Diagnosis of ALD - the diagnosis of ALD can be made by either biochemical or molecular/genetic evidence (plasma VLCFA or ABCD1 mutation analysis) supportive of ALD as the cause of cerebral demyelination
* Evidence of active cerebral disease - defined as the presence of gadolinium enhancement on a single brain MRI study - MRI used for eligibility determination may be performed at an outside institution; the most recent MRI used to determine eligibility must be within 2 calendar months of the date of enrollment on this study
* ALD MRI (Loes) score ≥ 10
* Off of N-acetylcysteine, systemic immunosuppressive drugs or any other therapeutic intervention (except hydrocortisone and/or fludracortisone for the treatment of adrenal insufficiency) for ≥ 10 days prior to the first IT-MSC dose
* Life expectancy of >6 months as determined by the enrolling researcher and documented in the medical record
* Voluntary written consent provided by parent(s)/guardian(s)

Exclusion Criteria:

* A candidate for allogeneic hematopoietic stem cell transplantation as determined by the University of Minnesota Inherited Metabolic and Storage Disease group
* Inability to undergo sedation, lumbar puncture or MRI studies for any reason
* Inability to stay in Minnesota for therapy through the day 28 evaluation

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Day 28 post intrathecal injection of MSC
  Determine the maximum tolerated dose (MTD) of intrathecally-administered allogeneic, third-party mesenchymal stem cells (IT-MSC) in patients with active, advanced cerebral adrenoleukodystrophy (cALD).

SECONDARY OUTCOMES:
Radiographic Response | 6 months
  Evaluate the incidence of, and time to, radiographic response in patients receiving IT-MSC for active, advanced cerebral adrenoleukodystrophy. Radiographic response is defined as the resolution of intravenous gadolinium contrast enhancement on brain MRI, or the absence of an increase in Loes score between the enrollment MRI and 6 month MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota